CLINICAL TRIAL: NCT04425291
Title: A Randomized, Double-Blind and Positive-Controlled Phase 3 Study to Evaluate the Immunogenicity and Safety of the 4-valent Human Papillomavirus (Types 6, 11, 16, 18) Recombinant Vaccine (Hansenula Polymorpha) and 9-valent Human Papillomavirus (Types 6, 11, 16, 18,31,33,45,52 and 58) Recombinant Vaccine (Hansenula Polymorpha) in Chinese Female Subjects Aged 20-45 Years
Brief Title: Evaluate the Immunogenicity and Safety of 4-valent and 9-valent HPV Recombinant Vaccine in Chinese Healthy Females
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Bovax Biotechnology Co., Ltd. (Industry)
Collaborators: Chongqing Bovax Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 4-HPV-3001
Record Dates: First submitted 2020-06-08; First posted 2020-06-11 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Cervical Cancer; Vulvar Cancer; Vaginal Cancer; CIN1; CIN2; CIN3; VaIN1; VaIN2; VaIN3; Genital Wart; VIN 1; VIN 2; VIN 3; AIS
MeSH Terms: conditions — Uterine Cervical Neoplasms; Vulvar Neoplasms; Vaginal Neoplasms; Condylomata Acuminata | interventions — Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 4-valent HPV Vaccine (Experimental): Participants in this arm would receive 4-valent Human Papillomavirus (Types 6, 11, 16 and18) Recombinant Vaccine (Hansenula Polymorpha)
  Interventions: Biological: 4-valent HPV Vaccine
- 9-valent HPV Vaccine (Experimental): Participants in this arm would receive 9-valent Human Papillomavirus (Types 6, 11, 16, 18,31,33,45,52 and 58) Recombinant Vaccine (Hansenula Polymorpha)
  Interventions: Biological: 9-valent HPV Vaccine
- GARDASIL® (Active Comparator): Participants in this arm would receive GARDASIL®
  Interventions: Biological: GARDASIL®

INTERVENTIONS:
Biological: 4-valent HPV Vaccine — Subjects received 3 doses of 4-valent HPV vaccine according to a 0, 2, 6-month schedule.
  Arms: 4-valent HPV Vaccine
Biological: 9-valent HPV Vaccine — Subjects received 3 doses of 9-valent HPV vaccine according to a 0, 2, 6-month schedule.
  Arms: 9-valent HPV Vaccine
Biological: GARDASIL® — Subjects received 3 doses of GARDASIL® according to a 0, 2, 6-month schedule.
  Arms: GARDASIL®

SUMMARY:
The study will evaluate the immunogenicity and safety of 4-valent and 9-valent HPV recombinant vaccine in Chinese healthy females 20 to 45 years of age.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese women aged 20-45 who can provide legal identification;
2. The subject agreed to participate in the study, and voluntarily signs the informed consent;
3. Subjects are able to understand the study procedures and participate in follow-up according to the study requirements;
4. When the subjects were enrolled, the urine pregnancy test was negative, they were not in the lactation period and had no family planning within 7 months after enrollment.2 weeks before included in the study, effective contraceptive measures has been adopted and agreed to in the first seven months after the study (vaccinations after 1 months ago) continue to adopt effective contraceptive measures (effective contraceptive measures including the pill or condoms, etc );

Exclusion Criteria:

1. Have been vaccinated with commercially available HPV vaccine in the past or planned to be vaccinated with commercially available HPV vaccine during the study period;Or have participated in a clinical trial of the HPV vaccine;
2. Has a history of cervical diseases, such as cervical screening showing abnormal results including CIN or a history of hysterectomy (vaginal or total abdominal hysterectomy) or pelvic radiation therapy. Has a history of genital diseases (such as vulvar intraepithelial neoplasia, vaginal intraepithelial neoplasia, genital warts, vulvar cancer, vaginal cancer and anal cancer, etc.) or has a previous sexual history (including syphilis, gonorrhea, chancre, venereal lymphatic granuloma, granuloma inguinal);
3. A history of severe allergies requiring medical intervention, such as anaphylactic shock, anaphylactic laryngeal edema, allergic purpura, thrombocytopenic purpura, local allergic necrosis reaction (Arthus reaction), etc;
4. Have an acute illness or an acute episode of a chronic illness within 3 days prior to vaccination or the use of antipyretic, analgesic and antiallergic drugs (e.g., acetaminophen, ibuprofen, aspirin, loratadine, cetirizine, etc.);
5. Subjects received inactivated or recombinant vaccines within 14 days prior to study enrollment, or attenuated live vaccines within 28 days prior to study enrollment;
6. Subjects present with immune impairment or have been diagnosed with congenital or acquired immune deficiency, HIV infection, lymphoma, leukemia, systemic lupus erythematosus (SLE), rheumatoid arthritis, juvenile rheumatoid arthritis (JRA), inflammatory bowel disease or other autoimmune diseases. Long-term immunosuppressive therapy, e.g., long-term (more than 2 weeks) treatment with glucocorticoids (e.g., prednisone or similar drugs);
7. Has been diagnosed with a severe congenital malformation or chronic disease such as Down syndrome, heart disease, liver disease, kidney disease, diabetes, etc., which may interfere with the conduct or completion of the study;
8. Subject receives any immunoglobulin or blood product within 3 months prior to the first dose of vaccination;
9. Participating in other (drug or vaccine) clinical trials prior to enrollment or planning to participate during the study;
10. Has been diagnosed with an infectious disease, such as tuberculosis, viral hepatitis and/or HIV infection;
11. A history or family history of convulsions, epilepsy, encephalopathy and mental illness;
12. Have contraindications to intramuscular injection, such as having been diagnosed with thrombocytopenia, any coagulation disorder or receiving anticoagulant therapy;
13. Absence of a spleen, functional absence of a spleen, and absence or removal of a spleen in any case;
14. Body temperature ≥37.3℃ (underarm body temperature);
15. Subjects may be unable to comply with the study procedure, comply with the agreement, or plan to permanently relocate from the region prior to completion of the study, or may be permanently absent from the region during the scheduled visit;
16. In the opinion of the investigators, the subjects had any other factors that made them unsuitable to participate in the clinical trial.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1680 (Actual)
Dates: Start 2020-05-28 (Actual); Primary Completion 2021-09-06 (Actual); Study Completion 2021-09-06 (Actual)

PRIMARY OUTCOMES:
Percentage of participants 20 to 45 Years of Age that achieve the neutralizing antibody serostatus cutoffs for seroconversion to HPV Types 6, 11, 16 and 18 at least 1 month post Dose 3. | 1 month post vaccination 3 (Month 7)

SECONDARY OUTCOMES:
The neutralizing antibody GMTs for HPV Types 6, 11, 16 and 18 in participants 20 to 45 Years of Age at least 1 month post Dose 3. | 1 month post vaccination 3 (Month 7)
Percentage of participants that achieve neutralizing antibody quadruple growth ratefor HPV Types 6, 11, 16 and 18 in participants 20 to 45 Years of Age at least 1 month post Dose 3. | 1 month post vaccination 3 (Month 7)
Percentage of participants that achieve neutralizing antibody quadruple growth rate or achieve the neutralizing antibody serostatus cutoffs for HPV Types 6, 11, 16 and 18 in participants 20 to 45 Years of Age at least 1 month post Dose 3. | 1 month post vaccination 3 (Month 7)
The neutralizing antibody GMTs for HPV Types 31, 33, 45 and 52 in participants 20 to 45 Years of Age at least 1 month post Dose 3. | 1 month post vaccination 3 (Month 7)
Percentage of participants that achieve neutralizing antibody quadruple growth ratefor HPV Types 31, 33, 45 and 52 in participants 20 to 45 Years of Age at least 1 month post Dose 3. | 1 month post vaccination 3 (Month 7)
Percentage of participants that achieve neutralizing antibody quadruple growth rate or achieve the neutralizing antibody serostatus cutoffs for HPV Types 31, 33, 45 and 52 in participants 20 to 45 Years of Age at least 1 month post Dose 3. | 1 month post vaccination 3 (Month 7)
Percentage of Participants Who Report at Least 1 Solicited Injection-site and Systemic Adverse Event 30 minutes post any vaccination | 30 minutes post any vaccination
Percentage of Participants Who Report at Least 1 Solicited Adverse Event 7 days post any vaccination | 7 days post any vaccination
Percentage of Participants Who Report at Least 1 Solicited and Unsolicited Adverse Event 30 days post any vaccination | 30 days post any vaccination
Percentage of Participants Who Experience at Least 1 Serious Adverse Event (SAE) from 1st vaccination to the completion of study | Day 1 to 6 months post vaccination 3
Percentage of Participants Who Experience Pregnancy from 1st vaccination to the completion of study | Day 1 to 6 months post vaccination 3

CONTACTS AND LOCATIONS:
Locations (1):
- Yangchun Center For Disease Prevention And Control, Yangchun, Guangdong, China

IPD SHARING:
Plan to Share IPD: No